CLINICAL TRIAL: NCT02898610
Title: CONVINCE - (COlchicine for preventioN of Vascular Inflammation in Non- CardioEmbolic Stroke) - a Randomised Clinical Trial of Low-dose Colchicine for Secondary Prevention After Stroke
Brief Title: Colchicine for Prevention of Vascular Inflammation in Non-cardio Embolic Stroke
Acronym: CONVINCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Health Research Board, Ireland (Other); Irish Heart Foundation (Other); University of Limerick (Other); University of Edinburgh (Other); National University of Ireland, Galway, Ireland (Other); Universitat de Lleida (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-004505-16
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Attack, Transient; Stroke
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine treatment (Active Comparator): Colchicine 0.5mg/day plus usual care for 60 months
  Interventions: Drug: Colchicine
- Usual Standard of care alone (No Intervention): Normal standard of care remains for these patients

INTERVENTIONS:
Drug: Colchicine
  Arms: Colchicine treatment

SUMMARY:
This study evaluates the use of Colchicine in adults over 40 years of age who have suffered an ischaemic stroke or transient ischaemic attack NOT caused by cardiac embolism or other defined causes. Patients will be randomised to 0.5 mg/day of Colchicine plus usual care, or to usual care alone.

To investigate the efficacy of low dose colchicine (0.5mg/day) plus usual care (defined as antiplatelet, lipid-lowering, antihypertensive treatment, and appropriate lifestyle advice) compared with usual care alone to prevent non-fatal recurrent ischaemic stroke, myocardial infarction, cardiac arrest, hospitalization for unstable angina and vascular death after ischaemic stroke or transient ischaemic attack (TIA) not caused by cardiac embolism or other defined causes unrelated to atherosclerosis

DETAILED DESCRIPTION:
Inflammation is a key pathophysiological contributor to unstable atherosclerotic plaque and thrombo-embolic events, stroke, myocardial infarction, and vascular death. Internationally, clinical trials are targeting atherosclerotic inflammation in patients with coronary disease using methotrexate, colchicine, and canukinumab.

Aims:

The primary aim is to compare low-dose colchicine (0.5mg/day) plus usual care, to usual care alone, to prevent non-fatal recurrent ischaemic stroke and coronary events and vascular death after non-severe, noncardioembolic TIA/stroke. Secondary objectives will investigate safety of low-dose colchicine, and efficacy for each component of the primary outcome, fatal and non-fatal events, disabling and non-disabling stroke, effect modification by prespecified subgroups, and impact on direct health care costs, adjusted for quality-adjusted life years.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent consistent with ICH-GCP guidelines and local laws signed prior to all trial-related procedures.
2. Age 40 years or greater
3. Either,

   * ischaemic stroke without major disability (modified Rankin score 3 or less)
   * or high-risk TIA
4. Qualifying stroke/TIA probably caused by large artery stenosis, small artery occlusion (lacunar stroke), or cryptogenic embolism, with cardiac embolism or other defined stroke mechanism deemed unlikely in the opinion of the treating physician.
5. GFRgreater than or equal to 50 ml/min.
6. In the opinion of the treating physician, patient is medically-stable, capable of participating in a randomised trial, and willing to attend follow-up.

Exclusion Criteria:

1. Cardio-embolic stroke/TIA, probably caused by identified atrial fibrillation (permanent or paroxysmal), in the opinion of the treating physician.
2. Cardio-embolic stroke/TIA probably caused by other identified cardiac source (intra-cardiac thrombus, endocarditis, metallic heart valve, low ejection fraction <30%), in the opinion of the treating physician.
3. Stroke/TIA caused by dissection, endocarditis, paradoxical embolism, drug use, venous thrombosis, within 48 hours aftercarotid or cardiac surgery, hypercoagulability states, migraine, or inherited cerebrovascular disorders (eg. Fabry's disease, CADASIL), in the opinion of the treating physician.
4. History of myopathy or myalgias with raised creatine kinase (CK) on statin therapy.
5. Blood dyscrasia defined as anaemia (haemoglobin <10g/dL), thrombocytopenia (platelet count <150 x109/L) or leucopenia (white cell count <4 x109/L) at randomisation.
6. Impaired hepatic function (transaminases greater than twice upper limit of normal) at randomisation.
7. Concurrent treatment with moderate or strong CYP3A4 inhibitors (clarithromycin, erythromycin, telithromycin, other macrolide antibiotics, ketoconazole, itraconazole, voriconazole, ritonavir, atazanavir, indinavir, other HIV protease inhibitors, verapamil, diltiazem, quinidine, digoxin, disulfiram) or P-gp inhibitors (cyclosporine) at randomisation.
8. Symptomatic peripheral neuropathy and pre-existing progressive neuromuscular disease
9. Inflammatory bowel disease (Crohn's or ulcerative colitis) or chronic diarrhoea.

9. Dementia, sufficient to impair independence in basic activities of daily living.

10. Active malignancy, known hepatitis B or C, or HIV infection prior to qualifying stroke/TIA.

11. Impaired swallow preventing oral administration of study medication. 12. History of poor medication compliance. 13. Unlikely to comply with study procedures and follow-up visits due to severe or fatal comorbid illness or other factor (eg. inability to travel for follow up visits), in opinion of randomising physician.

14. Pregnancy, breast-feeding, or pre-menopausal women 15. Patient concurrently participating in another clinical trial with an investigational drug or device, or use of investigational drug within 30 days or 5 half-lives before the Screening visit (whichever is longer) 16. Known allergy or sensitivity to colchicine.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3154 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Recurrence of non-fatal ischemic stroke | any time within 60 month
  Any recurrence of non-fatal ischemic stroke
on-fatal Major Cardiac event | any time within 60 months
  Non-fatal hospitalization for unstable angina, myocardial infarction, cardiac arrest
Vascular death | 60 months
  Fatal ischemic stroke, myocardial infarction, cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Prof Peter Kelly, Study Director — Mater Hospital
Locations (145):
- Belgium (11):
  - Uza, Antwerpen, Antwerp
  - AZ Sint Jan, Bruges
  - AZ St. Lucas, BRUGGE, Bruges
  - UCL, Brussels, Brussels
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
  - AZ Groeninge Kortrijk, Kortrijk
  - UZ Leuven, Leuven
  - CHC Liege, Liège
  - AZ Damiaan, OOSTENDE, Ostend
  - AZ Delta, ROESELARE, Roeselare
- Canada (3):
  - Foothills Medical Centre, Calgary, Calgary
  - Kingston Hospital, Kingston
  - Vancouver General Hospital, Vancouver
- Czechia (2):
  - St. Anne´s University Hospital, Brno
  - Hospital Jihlava, Jihlava
- Denmark (4):
  - Bispebjerg Hospital, Bispebjerg
  - Rigshospitalet Glostrup, Glostrup Municipality
  - Herlev Hospital, Herlev
  - Nordsjællands Hospital, Hillerød
- Tartu University Hospital, Tartu, Estonia
- Germany (23):
  - Rhön-Klinikum Campus Bad Neustadt, Bad Neustadt an der Saale
  - Vivantes Auguste-Viktoria Klinikum, Berlin
  - Vivantes Humboldt-Klinikum, Berlin
  - Vivantes Klinikum Neukölln, Berlin, Berlin
  - St. Josef-Hospital Klinikum der Ruhr-Universität Bochum, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Krankenhaus Buchholz, Buchholz
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitätsklinikum Essen, Essen
  - Frankfurt University Hospital, Frankfurt
  - Klinikum Fulda gAG, Universitätsmedizin Marburg-Campus Fulda, Fulda
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Krakenhaus Martha Maria Halle Dolau, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Klinikum Main-Spessart, Standort Krankenhaus Lohr, Lohr
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Klinikum der Universität München, München
  - Mediclin-Fachklinik Rhein/Ruhr, Rheine
  - Medinos Kliniken des Landkreises Sonneberg, Sonneberg
  - Universitätsklinikum Würzburg, Würzburg
- Ireland (15):
  - Cavan General Hospital, Cavan, Cavan
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Connolly Hospital, Blanchardstown, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St James's Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - Tallaght University Hospital, Dublin
  - Galway University Hospital, Galway
  - St Lukes General Hospital, Kilkenny
  - University Hospital Limerick, Limerick
  - Our Lady of Lourdes, Drogheda, Louth
  - Sligo University Hospital, Sligo
  - South Tipperary General Hospital, Clonmel, Tipperary
  - University Hospital Waterford, Waterford
- Lithuania (2):
  - Lithuanian University Hospital of Health Sciences Kaunos Klinikos, Kaunas
  - Vilnius University Hospital Santaros Clinics, Vilnius
- Netherlands (4):
  - Academic Medical Center, Amsterdam
  - Gelre Ziekenhuis Apeldoorn, Apeldoorn
  - Reinier de Graaf Hospital, Delft
  - Radboud University Medical Centre, Nijmegen
- Poland (4):
  - Hospital Nicholas Copernicus, Gdansk
  - Specialist Hospital of Saint Luke, Gmina Końskie
  - Medical University of Silesia Hospital No7, Rokietnica
  - Institute of Psychiatry and Neurology, Warsaw
- Portugal (3):
  - Hospital de Santa Maria, Centro Hospitalar Lisboa Norte, Lisbon
  - Hospital Egas Moniz, Lisbon
  - Hospital Universitario de Sao Jao, Porto
- Spain (13):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - H. de Albacete, Albacete
  - Hospital de Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Moises Broggi. Comprehensive Health Consortium, Barcelona
  - H U. Josep Trueta, Girona, Girona
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - H. U. Ramón y Cajal, Madrid, Madrid
  - Centro Medico de Asturias, Oviedo
  - H Parc Taulí de Sabadell, Sabadell
  - H U. Virgen del Rocío, Sevilla, Seville
  - Hospital Virgen Macarena Sevilla, Seville
  - H Joan XXIII, Tarragona, Tarragona
- University Hospital Bern, Bern, Switzerland
- United Kingdom (59):
  - Bronglais General Hospital, Aberystwyth
  - Aintree University Hospital, Aintree
  - Monklands Hospital, Airdrie
  - Antrim Area Hospital, Antrim
  - William Harvey Hospital, Ashford
  - Royal Victoria Hospital, Belfast
  - Royal Blackburn Hospital, Blackburn
  - Pilgrim Hospital, Boston
  - Royal Bournemouth Hospital, Bournemouth
  - West Suffolk Hospital, Bury St Edmunds
  - Addenbrookes Hospital, Cambridge
  - Kent and Canterbury Hospital, Canterbury
  - Countess of Chester Hospital, Chester
  - Chesterfield Royal Hospital, Chesterfield
  - St Richards Hospital, Chichester
  - Craigavon Area Hospital, Craigavon
  - Northumbria Specialist Emergency Care Hospital, Cramlington
  - Croydon University Hospital, Croydon
  - Royal Derby Hospital, Derby
  - North Durham University Hospital, Durham
  - South West Acute Hospital, Enniskillen
  - Royal Devon & Exeter Hospital, Exeter
  - Queen Elizabeth Hospital Gateshead, Gateshead
  - Medway Maritime Hospital, Gillingham
  - Hairmyres Hospital, Glasgow
  - Queen Elizabeth University Hospital Glasgow, Glasgow
  - Wycombe Hospital, High Wycombe
  - Raigmore Hospital, Inverness
  - Kingston Hospital, Kingston
  - Leicester Royal Infirmary, Leicester
  - University Hospital Lewisham, Lewisham
  - Lincoln County Hospital, Lincoln
  - Royal Liverpool University Hospital, Liverpool
  - Charing Cross Hospital, London
  - King's College Hospital, London
  - Royal London Hospital, London
  - St George's Hospital, London
  - St Thomas' Hospital, London
  - University College London Hospital, London
  - Altnagelvin Area Hospital, Londonderry
  - Luton & Dunstable University Hospital, Luton
  - Queen Elizabeth the Queen Mother Hospital, Margate
  - Norfolk and Norwich Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Peterborough Hospital, Peterborough
  - Derriford Hospital, Plymouth
  - Royal Hallamshire Hospital, Sheffield
  - Southend University Hospital, Southend
  - Stepping Hill Hospital, Stockport
  - Royal Stoke University Hospital, Stoke
  - Sunderland Royal Hospital, Sunderland
  - King's Mill Hospital, Sutton in Ashfield
  - Great Western Hospital, Swindon
  - Princess Royal Hospital, Telford
  - Royal Cornwall Hospital, Truro
  - Whiston Hospital, Whiston
  - New Cross Hospital, Wolverhampton
  - Worthing Hospital, Worthing
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: Yes
A summary report of the trial will be provided to the Ethics Committees and relevant Regulatory Authority within as per national legal requirements in participating countries
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within one year

REFERENCES:
- [Background] Kelly P, Lemmens R, Weimar C, Walsh C, Purroy F, Barber M, Collins R, Cronin S, Czlonkowska A, Desfontaines P, De Pauw A, Evans NR, Fischer U, Fonseca C, Forbes J, Hill MD, Jatuzis D, Korv J, Kraft P, Kruuse C, Lynch C, McCabe D, Mikulik R, Murphy S, Nederkoorn P, O'Donnell M, Sandercock P, Schroeder B, Shim G, Tobin K, Williams DJ, Price C. Long-term colchicine for the prevention of vascular recurrent events in non-cardioembolic stroke (CONVINCE): a randomised controlled trial. Lancet. 2024 Jul 13;404(10448):125-133. doi: 10.1016/S0140-6736(24)00968-1. Epub 2024 Jun 7. PMID 38857611
- [Derived] Maes L, Walsh C, Weimar C, Purroy F, Price C, Clarke B, Castro P, Czlonkowska A, Cuadrado-Godia E, Fischer U, Fonseca AC, Hill MD, Jatuzis D, Korv J, Kruuse C, Mikulik R, Nederkoorn PJ, Sztriha L, Thieme M, Kelly P, Lemmens R. Effect of colchicine for secondary prevention according to stroke subtype: A secondary analysis of the CONVINCE randomized trial. Int J Stroke. 2025 Dec 2:17474930251406818. doi: 10.1177/17474930251406818. Online ahead of print. PMID 41328787
- [Derived] Akl E, Sahami N, Labos C, Genest J, Zgheib A, Piazza N, Jolly S. Meta-Analysis of Randomized Trials: Efficacy and Safety of Colchicine for Secondary Prevention of Cardiovascular Disease. J Interv Cardiol. 2024 Mar 12;2024:8646351. doi: 10.1155/2024/8646351. eCollection 2024. PMID 38505729
- [Derived] Bouabdallaoui N, Tardif JC. Colchicine in the Management of Acute and Chronic Coronary Artery Disease. Curr Cardiol Rep. 2021 Jul 16;23(9):120. doi: 10.1007/s11886-021-01560-w. PMID 34269908